CLINICAL TRIAL: NCT03392519
Title: Functional Magnetic Resonance Imaging and Diffusion Tensor Imaging Study About Reorganization and Recovery Mechanism of Brain Neural Network for Chronic Stroke Patients
Brief Title: Brain Imaging Study of Brain Plasticity in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-07-082
Record Dates: First submitted 2017-12-25; First posted 2018-01-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2019-09

CONDITIONS: Chronic Stroke
Keywords: Brain connectivity; Magnetic resonance imaging; Brain plasticity; Recovery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic stroke: More than 3 months post-stroke Ischemic or hemorrhagic stroke
  Interventions: Other: Chronic stroke

INTERVENTIONS:
Other: Chronic stroke — MRI data acquisition and behavioral test

SUMMARY:
In chronic stroke patients, brain network reorganization and recovery mechanism are investigated after stroke onset using functional MRI and diffusion tensor imaging analyses.

ELIGIBILITY:
Inclusion Criteria:

* more than 3 months post-stroke
* ischemic or hemorrhagic stroke
* a person who understands the experiment and has a willingness to participate and signs the agreement

Exclusion Criteria:

* User of artificial heartbeat
* Patients with claustrophobia
* Patients with metal implants
* Patients who are contraindicated for other common MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A person who was inpatient at subacute stage at the Samsung Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between strength of connection and the Fugl-Meyer Assessment score | Through study completion, an average of 1 year
  Strength of connection is obtained by calculating a correlation coefficient between time courses of both regions in fMRI data.
Correlation coefficient between the FA value of a tract and the Fugl-Meyer Assessment score | Through study completion, an average of 1 year
  FA value is obtained by assessing a diffusion anisotropy of a specific tract in DTI data.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No